CLINICAL TRIAL: NCT04057313
Title: Coffee Intake in HemoDialysis and Headache (CoffeeHD): a Randomized Double Blind Multicenter Clinical Trial
Brief Title: Coffee in Hemodialysis and Headache
Acronym: CoffeeHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Mabel Aoun, Dr, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CoffeeHD2019
Record Dates: First submitted 2019-08-11; First posted 2019-08-15 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Hemodialysis Complication
Keywords: Coffee; Headache; Intra-dialytic hypotension
MeSH Terms: conditions — Headache | interventions — Coffee

STUDY DESIGN:
Intervention Model Description: A randomized multicenter trial: hemodialysis patients in three dialysis units will be randomized to two groups, group 1 will take coffee for 4 weeks, group 2 will take decaffeinated coffee for 4 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will be ensured by an outsider who will hold the coffee cups to nurses with the name of patients on the cups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Group 1 will receive 80 cc of coffee in the dialysis session
  Interventions: Dietary Supplement: Coffee
- Group 2 (Placebo Comparator): Group 2 will receive 80 cc of decaffeinated coffee in the dialysis session
  Interventions: Dietary Supplement: Coffee

INTERVENTIONS:
Dietary Supplement: Coffee — Coffee used will be the boiled unfiltered Arabica coffee

SUMMARY:
Coffee is the most consumed drink worldwide, sometimes needed to boost energy and other times to entertain social connectivity. Caffeine is mostly present unbound in the plasma, only 10 to 30% of caffeine binds to plasma proteins. It is distributed freely into the intracellular space, and it has a small distribution volume. Therefore, caffeine can pass through the dialysis membrane during a standard hemodialysis session. In hemodialysis patients, headache occurs in 40 to 75% of patients. Some authors have suggested that one of the reasons of headache during hemodialysis is caffeine withdrawal. This trial aims to find whether coffee intake during hemodialysis reduces the headache episodes. It is a randomized double blind multicenter trial where 160 patients will be randomized to 2 groups: group 1 of 80 patients will be given a cup of coffee each dialysis session for 4 weeks and group 2 will receive decaffeinated coffee each dialysis session for 4 weeks.

DETAILED DESCRIPTION:
Coffee is the most consumed drink worldwide, sometimes needed to boost energy and other times to entertain social connectivity. It is known also to cause addiction and thus be a cause for withdrawal symptoms such as headache and irritability. Coffee is not contra-indicated in patients with chronic kidney disease. Caffeine is mostly present unbound in the plasma, only 10 to 30% of caffeine binds to plasma proteins. It is distributed freely into the intracellular space, and it has a small distribution volume within the body around 0,7L/kg. Therefore, caffeine can pass through the dialysis membrane during a standard hemodialysis session. In hemodialysis patients, intra-dialytic hypotension, fatigue post-dialysis and headache occur in 40 to 75% of patients. Some authors have suggested that one of the reasons of headache during hemodialysis is caffeine withdrawal.

This trial aims to find out whether coffee consumption during dialysis could decrease headache episodes.

Methods

Study setting All patients on chronic hemodialysis in three Lebanese dialysis units, Saint-Georges Ajaltoun hospital, Hôtel-Dieu de France and Bellevue Medical Center will be included.

Trial design and participants This is a randomized, controlled, double-blind, multi-center clinical trial. Patients will be randomized to one of two arms and then group one will receive the coffee during hemodialysis session and group two will receive decaffeinated coffee.

Blinding will be ensured by designating an external employee that will hold the cups of coffee to the unit's nurses every day with the name of each patient on the cup.

Randomization Patients will be assigned to receive coffee during hemodialysis or not using a 1:1 allocation ratio.

Interventions Patients will be randomly assigned to one of two groups: Group 1 will receive a cup of coffee (80 cc) in the middle of the dialysis session every session for 4 weeks. Group 2 will receive non-caffeinated cup of coffee (80 cc) in the middle of the dialysis session every session for 4 weeks. The coffee that will be used is the boiled unfiltered Arabica coffee with a ratio of water to coffee of 800 ml/125 g. Patients can add sugar to their coffee if they want. Ultrafiltration rate will not exceed 13 mL//kg/hour for all included patients.

Participant timeline Every patient will be followed from first day of randomization till the end of the month (4 weeks follow-up).

Sample size calculation If we consider a two-sided alpha of 5% and power of 90% and a prevalence of headache in the dialysis population up to 75% that will be reduced by 25% in the group taking caffeine, the total sample size needed would be 160 patients, 80 in each arm.

Data collection

Variables that will be collected include:

* Personal information: age, sex, smoking, alcohol intake per week, hypertension (at least one antihypertensive drug)
* Caffeine intake: number of coffee cups at home per day (outside the dialysis session), coffee intake before the dialysis session (yes/no), coffee intake during the dialysis session (yes/no)
* Medical history: diabetes, hypertension, coronary artery disease, history of headache or migraine
* Medications: beta blockers, antidepressants, benzodiazepine
* Dialysis sessions related information: dialysis vintage (months), urea reduction ratio (URR) of the month
* Clinical variables: number of intra-dialytic hypotensive the month before the trial and during the trial, number of intra-dialytic and home headache episodes during the trial, pre-dialysis systolic and diastolic blood pressure and heart rate of the first and the last session of the trial, insomnia before and at the end of the trial, energy after a dialysis session before and after the trial and irritability before and after the trial.
* Adverse events will be also reported such as arrhythmia, tachycardia or hypertension.

Statistical analysis Continuous variables will be presented as mean ± standard deviation (SD) and categorical variables as percentages. The effectiveness of the randomization will be checked by comparing baseline variables with the appropriate tests.

The analysis will depend on the distribution of the outcome variables:

If outcome variables are normally or quasi-normally distributed, Hotelling's T-Squared will be used as an overall multivariate test for the difference between the 2 groups, followed by t-tests to assess individual outcomes.

If outcome variables are skewed, the Mann-Whitney test will be used. Bonferroni correction will be used to adjust for multiple comparisons. A P-value of ≤0.05 is considered statistically significant.

Definitions Hypotensive episodes are defined as drop of systolic blood pressure below 90 mmHg or of 20 mmHg accompanied with clinical symptoms such as muscle cramps, chest pain, dyspnea, dizziness, headache, abdominal pain, nausea, vomiting, weakness, anxiety, paleness and sweating. Hypotensive episodes during dialysis usually occur in 15-30% of cases.

Irritability and energy will be assessed based on two questions:

* Have you been a very nervous person, irritated by minor incidents? (yes/no)
* How much energy do you feel after your dialysis session on a scale from 1 to 10?

Insomnia will be assessed by two questions: have you any difficulty sleeping at night? (yes/no), how many hours do you sleep at night?

Ethical approval The study will get approval from the ethics committee of Saint-Joseph University and is in agreement with the Helsinki Declaration of 1975.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients > 18 years old on chronic hemodialysis

Exclusion Criteria:

* patients with a history of chronic or paroxysmal atrial fibrillation
* patients on chronic systematic pain killers
* patients with a problem of swallowing food or drinks
* patients who are coffee allergic or intolerant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
number of headache episodes | 4 weeks
  number of headache episodes during or immediately after dialysis over 12

SECONDARY OUTCOMES:
number of intra-dialytic hypotensive episodes | 4 weeks
  number of intra-dialytic hypotensive episodes during trial over 12
number of sleeping hours per night | 4 weeks
  number of sleeping hours per night during the trial (average)
energy after dialysis | 4 weeks
  energy after dialysis on a scale from 1 to 10 (1 is no energy and 10 is full energy)
irritability | 4 weeks
  irritability during the trial (question: are you easily irritated? yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Mabel Aoun, MD, Principal Investigator — Saint-Joseph University
Locations (1):
- Saint-Georges Hospital, Ajaltoun, Kesrouan, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aoun MH, Hilal N, Beaini C, Sleilaty G, Hajal J, Boueri C, Chelala D. Effects of Caffeinated and Decaffeinated Coffee on Hemodialysis-Related Headache (CoffeeHD): A Randomized Multicenter Clinical Trial. J Ren Nutr. 2021 Nov;31(6):648-660. doi: 10.1053/j.jrn.2021.01.025. Epub 2021 Mar 12. PMID 33715955